CLINICAL TRIAL: NCT01582542
Title: Usage of Desmopressin fo Improving Nocturnal Enuresis in Patients After Radical Cystectomy With Orthotopic Bladder Reconstruction
Brief Title: Desmopressin for Improving Nocturnal Enuresis in Patients After Radical Cystectomy With Bladder Reconstruction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0366-11-RMC
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Desmopressin (Experimental)
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Patients after radical cystectomy with orthotopic bladder reconstruction that suffer from night time urinary incontinence will be enrolled in the study. They will be given for a period of one month after informed consent, Desmopressin At a dosage of 0.1 M"G per day. The rate of improvement of night time urinary incontinence will be measured.
  Other Names: Minerine; Nocturnal Enuresis

SUMMARY:
The purpose of this study is to prospectively assess whether Desmopressin, given for a period of month to patients after radical cystectomy with orthotopic bladder reconstruction, improves and lowers the rate of nocturnal enuresis.

DETAILED DESCRIPTION:
We will prospectively assess the utilization of Desmopressin in improving nocturnal enuresis in patients after radical cystectomy with orthotopic bladder reconstruction.

Patients after radical cystectomy with neobladder reconstruction will be given Desmopressin 0.1 mg once a day for a duration of one month.

Before beginning treatment patients will be given the NNES-Q questionnaire to assess severity of nocturnal enuresis.

At the end of treatment, the same questionnaire will be given to all patients to assess if nocturnal enuresis improved.

Sodium levels will be tested before treatment, 2 weeks after beginning treatment and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Able to give informed consent
* Patients afte radical cystectomy with orthotopic bladder reconstruction with night time incontinence

Exclusion Criteria:

* Patients with after radical cystectomy with orthotopic bladder reconstruction with daytime urinary incontinence
* Patients already treated with Desmopressin due to other reasons.
* Patients with an allergy or insensitivity to Desmopressin.
* Patients with known hyponatremia
* Patients with severe chronic renal failure and creatinine clearance of below 50 cc/sec.
* Patients with severe congestive heart failure
* Patients with active urinary tract infection
* Patients taking drug therapy which can interact with Desmopressin and affect it's action.Examples include Diuretics, Tricyclic antidepressants, Carbamezapine and Chlorpropamide AND Indomethacin.
* Patients with an indwelling urinary catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Rate of improvement in Nocturnal incontinence | One month

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Yossepowitch, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Institute of Urology, Rabin Medical Cetner, Petah Tikva, Petach Tiqva, Israel